CLINICAL TRIAL: NCT04992013
Title: Genomically Guided Phase II Study to Evaluate the Clinical Benefit of Niraparib in Tumors Metastatic to the CNS
Brief Title: Niraparib in Tumors Metastatic to the CNS
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Principal Investigator, Priscilla Brastianos, Principal Investigator, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 21-154
Record Dates: First submitted 2021-07-28; First posted 2021-08-05 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Metastatic Cancer; Central Nervous System Cancer
Keywords: Metastatic Cancer; Central Nervous System Cancer
MeSH Terms: conditions — Neoplasm Metastasis; Central Nervous System Neoplasms | interventions — niraparib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Niraparib (Experimental): Participants will receive niraparib 1x daily for each 28 day study treatment cycle up to 2 years or until disease worsens or unacceptable side effects occur.
  Interventions: Drug: Niraparib

INTERVENTIONS:
Drug: Niraparib — Capsule taken by mouth
  Other Names: Zejula

SUMMARY:
This research is being done to see how effective the drug niraparib is against cancer that has metastasized to the central nervous system (CNS).

* This research study involves the study drug niraparib.

DETAILED DESCRIPTION:
This is a single arm open-label study designed to evaluate the efficacy and safety of niraparib in treating cancer that has metastasized to the central nervous system (CNS).

The U.S. Food and Drug Administration (FDA) has not approved niraparib for cancer metastasized to the central nervous system (CNS) but it has been approved for other uses.

Niraparib is a type of drug called a "PARP inhibitor", which blocks DNA (the genetic material of cells) damage from being repaired or may prevent damage from occurring in the first place. In cancer treatment, inhibiting PARP may help kill cancer cells by not allowing the cancer cells to repair its DNA damage or prevent DNA damage associated with your diagnosis from occurring.

The research study procedures include screening for eligibility and study treatment including evaluations and follow up visits.

Participants will receive the study drug for up to 2 years or until their disease worsens, they have unacceptable side effects, or they meet one of the criteria to be removed from the study. Participants will then be followed every 4 months for up to 2 years.

It is expected that about 20 people will take part in this research study.

GlaxoSmithKline, a pharmaceutical company, is supporting this research study by providing funding for the study, including the study drug.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have histologically or cytologically confirmed disease from any solid tumor.
* Patients must be asymptomatic or minimally symptomatic from CNS metastases for at least 7 days prior to initiation of study therapy. Minimal symptoms is defined as not requiring escalating doses of steroids or seizure medications for at least 7 days prior to initiation of study therapy.
* Participants must have measurable disease in the CNS, defined as at least one lesion that can be accurately measured in at least one dimension as ≥10 mm.
* Participants must have progressive CNS lesions, as defined by one of the following:

  * Patients may have multiple progressive CNS lesions, some of which have been treated by SRS or surgery. Patients are eligible if they have one or more un-treated (by surgery or SRS) progressive lesions that is measurable.
  * Patients have measurable residual or progressive lesions after surgery.
  * Patients who have had prior WBRT and/or SRS are eligible but there needs to be unequivocal evidence of progression of at least one lesion treated by radiation (e.g. tissue diagnosis). Biopsy can be considered for definitive diagnosis.
  * Patients who have previously been treated with systemic therapy for CNS metastases are eligible.
* Diagnosis of triple negative breast cancer or ovarian cancer, or any cancer histology with the presence of alteration in BRCA1, BRCA2, PARP metabolism, DNA repair pathways and HRD (homologous recombination deficiency) genes in the metastatic site as described in Section 9.2 using a CLIA-certified assay. Specific genetic changes in the HRD signature or DNA repair pathway include mutations in ATM, BAP1, BARD1, BRCA1, BRCA2, BRIP1, MRE11A, NBN, PALB2, RAD50, RAD51B, RAD51C, RAD51D, RAD54B, RAD54L, ATR, XRCC2, and XRCC3.
* Age > 18 years. The toxicity of niraparib in children is unknown.
* ECOG performance status ≤ 2 (Karnofsky ≥ 60, see Appendix A).
* Participants must have normal organ and marrow function as defined below:

  * leukocytes ≥3,000/mcL
  * absolute neutrophil count ≥1,500/mcL
  * platelets ≥100,000/mcL
  * hemoglobin ≥9g/dL
  * total bilirubin total bilirubin < 1.5 x institutional upper limit of normal OR > 1.5 x institutional upper limit of normal allowed if direct bilirubin is within normal range. Patients with Gilberts will be eligible if total bili < 3.
  * AST(SGOT)/ALT(SGPT) ≤2.5 × institutional upper limit of normal
  * creatinine clearance ≥30 mL/min/1.73 m2 using the Cockcrof-Gault equation.
  * baseline QTc <480ms
* Female participant has a negative urine or serum pregnancy test within 72 hours prior to taking study treatment if of childbearing potential and agrees to abstain from activities that could result in pregnancy from screening through 180 days after the last dose of study treatment, or is of nonchildbearing potential. Nonchildbearing potential is defined as follows (by other than medical reasons):

  * ≥45 years of age and has not had menses for >1 year
  * Patients who have been amenorrhoeic for <2 years without history of a hysterectomy and oo phorectomy must have a follicle stimulating hormone value in the postmenopausal range upon screening evaluation
  * Post-hysterectomy, post-bilateral oophorectomy, or post-tubal ligation. Documented hysterectomy or oophorectomy must be confirmed with medical records of the actual procedure or confirmed by an ultrasound. Tubal ligation must be confirmed with medical records of the actual procedure, otherwise the patient must be willing to use a highly effective barrier methods throughout the study, starting with the screening visit through 180 days after the last dose of study treatment. See Section 4.4 for a list of acceptable birth control methods. Information must be captured appropriately within the site's source documents. Note: Abstinence is acceptable if this is the established and preferred contraception for the patient.
* Participant must agree to not breastfeed during the study or for 30 days after the last dose of study treatment.
* Ability to understand and the willingness to sign a written informed consent document.
* Tissue from a prior craniotomy or biopsy for clinical genetic sequencing (at least one FFPE block or 15 unstained slides). If CNS tissue is not available, extracranial tissue can be used for sequencing. Patients previously assessed for genetic sequencing who meet requirements of section 9.2.1 do not need to have additional tissue available for prospective genetic screening.
* Patients with progressive extracranial disease will not be excluded.
* Participant must agree to not donate blood during the study or for 90 days after the last dose of study treatment.
* Stable dose of corticosteroids for at least 7 days.
* Patients are allowed to remain on letrozole, anastrozole, exemestane, tamoxifen, fulvestrant, trastuzumab, bisphosphonates, denosumab or ovarian suppression therapy
* Ability to swallow capsules

Exclusion Criteria:

* Prior treatment with PARP inhibitor.
* Participants who have had chemotherapy, immunotherapy or radiotherapy within 2 weeks prior to entering the study or those who have continuing or unresolved ≥grade 2 adverse events due to agents administered more than 2 weeks earlier (except for patients who will receive letrozole, anastrozole, exemestane, tamoxifen, fulvestrant, trastuzumab, bisphosphonates, denosumab or ovarian suppression therapy).
* Participant must not have had major surgery ≤ 3 weeks prior to initiating protocol therapy and participant must have recovered from any surgical effects.
* Must not have received investigational therapy ≤ 4 weeks, or within a time interval less than at least 5 half-lives of the investigational agent, whichever is shorter, prior initiating protocol therapy.
* Participant has had radiation therapy encompassing >20% of the bone marrow within 2 weeks; or any radiation therapy within 1 week prior to Day 1 of protocol therapy.

Participant must not have a known hypersensitivity to niraparib components or excipients.

* Participant must not have received a transfusion (platelets or red blood cells) ≤ 4 weeks prior to initiating protocol therapy.
* Participant must not have received colony stimulating factors (e.g., granulocyte colony-stimulating factor, granulocyte macrophage colony stimulating factor, or recombinant erythropoietin) within 4 weeks prior initiating protocol therapy.
* Participant has had any known Grade 3 or 4 anemia, neutropenia or thrombocytopenia due to prior chemotherapy that persisted > 4 weeks and was related to the most recent treatment.
* Participant must not have any known history of myelodysplastic syndrome (MDS) or acute myeloid leukemia (AML).
* Participant must not have a serious, uncontrolled medical disorder, nonmalignant systemic disease, or active, uncontrolled infection. Examples include, but are not limited to, uncontrolled ventricular arrhythmia, recent (within 90 days) myocardial infarction, uncontrolled major seizure disorder, unstable spinal cord compression, superior vena cava syndrome, or any psychiatric disorder that prohibits obtaining informed consent.
* Participant must not have had diagnosis, detection, or treatment of another type of cancer ≤ 2 years prior to initiating protocol therapy (except basal or squamous cell carcinoma of the skin and cervical cancer that has been definitively treated)
* Unable to undergo MRI scans.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-04-05 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
Intracranial Clinical benefit rate | 8 Weeks
  Assessed by RANO criteria for brain metastases

SECONDARY OUTCOMES:
Extracranial clinical benefit rate | Up to 2 years
  Assessed by RECIST and duration of response
Intracranial disease progression | Time to the first occurrence of intracranial disease progression, or death from any cause up to 2 years
  Assessed by cumulative incidence function (CIF), which estimates the marginal probability of each competing event via cause-specific hazards
Extracranial disease progression | Time to the first occurrence of extracranial disease progression, or death from any cause up to 2 years
  Assessed by cumulative incidence function (CIF), which estimates the marginal probability of each competing event via cause-specific hazards
Overall Survival Rate | Up to 2 years
  Summarized using Kaplan-Meier.
Number of Participants With Treatment-Related Adverse Events as Assessed by CTCAE Version 5.0 | Up to 2 years
  The number and proportion of adverse events, graded as defined by CTCAE version 5.0 will be will be summarized according to system organ class and/or preferred term, severity (based on CTCAE grade), type of adverse event, and relation to study treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Priscilla Brastianos, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital Cancer Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: [contact information for Sponsor Investigator or designee]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Partners Innovations team at http://www.partners.org/innovation